CLINICAL TRIAL: NCT05173571
Title: Home Comprehensive Therapeutic Support Program in Patients With Pulmonary Fibrosis
Brief Title: Homecare Integral Support Program for IPF Patients
Acronym: PSPi-IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Maria Molina, MD, PhD, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PR118/18
Record Dates: First submitted 2020-10-27; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Homecare patient support
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Physical Therapy Modalities; Nurses

STUDY DESIGN:
Intervention Model Description: Minimal intervention study, pre- and post- supportive care effects on quality of life
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional and physical activity program (Experimental): Homecare IPF patient educational, nutritional and physical activity training based on patient's needs
  Interventions: Combination Product: Comprehensive patient support program (educational, physiotherapy, nutritional, emotional)

INTERVENTIONS:
Combination Product: Comprehensive patient support program (educational, physiotherapy, nutritional, emotional) — Identification of patient needs and non-pharmacological holistic approach, including education, emotion and nutrition (nurse) and optimization of physical activity (respiratory physiotherapist)
  Other Names: Nurse and Respiratory Physiotherapist holistic plan

SUMMARY:
Homecare patient support program especially designed for covering IPF patient needs, implemented for 12 months, for improving quality of life

DETAILED DESCRIPTION:
The proposed comprehensive IPF home care programme consists of: 1) improving patient's quality of life (autonomy, activity, emotional well-being and symptoms), 2) reducing the number and severity of side effects associated with the anti-fibrotic drug, 3) reducing the number of hospitalisations attributable to the disease, and 4) providing a rapid response to any problem associated with the disease (after diagnosis or progression) that may cause distress or require early action.

ELIGIBILITY:
Inclusion Criteria:

* IPF patients with FVC > 50% and DLCO > 30%, in whom pharmacological treatment with nintedanib was started at least one month before the start of the programme.

Exclusion Criteria:

* Hospitalised patients or those who have been hospitalised in the previous month, due to any kind of respiratory exacerbation or due to any other respiratory cause.
* Patients who are under home care controls (PADES) as this implies an advanced stage of the disease (forced vital capacity [FVC] less than 50% and the diffusion capacity of the lungs for carbon monoxide [DLCO] less than 30%) or, patients thathave a lack of autonomy due to comorbidities or respiratory failure
* Patients diagnosed in incipient phase who have neither symptoms nor limitation in their usual activities.
* Patients who have suffered any other life-threatening disease in the last 2 years, such as cancer or uncontrolled ischaemic heart disease.
* Inability to understand the information given to the patient, relating to the legal aspects of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Qulity of life | 12 months
  K-BILD score (global and by domains)

CONTACTS AND LOCATIONS:
Locations (1):
- IDIBELL. University Hospital of Bellvitge, L'Hospitalet de Llobregat, Spain